CLINICAL TRIAL: NCT03914911
Title: In Vivo Smart Biopsy Device Protocol In Radiology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dune Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-10-001
Record Dates: First submitted 2018-11-28; First posted 2019-04-16 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Image Guided Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): The radiologist will perform a routine ultrasonic guided biopsy procedure using the Smart Biopsy Device, with the device readings not visible (i.e. the radiologist will be blinded to device readings)
  Interventions: Device: Smart Biopsy Device

INTERVENTIONS:
Device: Smart Biopsy Device — The radiologist will perform a routine ultrasonic guided biopsy procedure using the smart biopsy system, with the device readings not visible (i.e. the radiologist will be blinded to device readings)

SUMMARY:
This study is designed to demonstrate the feasibility of use of the Smart Biopsy Device in real clinical settings.

DETAILED DESCRIPTION:
This is a single arm, multicenter study. It will be conducted in 3 medical centers, in the breast-imaging unit during ultrasonic guided core needle biopsy procedures performed in women with abnormality in the breast.

The study duration is only during the biopsy procedure, and the follow up period is 2 -3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age
* Undergoing ultrasonic guided core needle biopsy procedure due to abnormality in the breast
* Signed Informed Consent Form

Exclusion Criteria:

* Concurrent infectious disease
* Pregnancy or breastfeeding
* Participating in any other investigational study for either drug or device which can influence collection of valid data under this study
* Implanted devices / Implants in the operated breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) Adverse events (AEs) | The subjects will be followed for a period of 2 -3 weeks following the biopsy procedure
  AEs will be documented during the biopsy procedure and SAEs will be followed up to 3 weeks after the biopsy procedure. Rates of adverse events such as bleeding, hematoma, infection and pain will be compared to adverse events for similar procedures published in the literature and anticipated in the product risk analysis.
Correlation between pathology results and device readings | 2-3 weeks following biopsy procedure
  Correlation between pathology results and device readings
Ergonomic Assessment of the Smart Biopsy Device | At the day of the biopsy procedure
  A questionnaire will be completed by the radiologist and applicable radiology lab staff to assess the ease of device assembly and handling properties. Each of the eight questions will use the same four point rating scale. At the end of the study the average and standard deviation will be calculated for each of the questions.

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Weisenberg, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center Campus Beilinson, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Dune Medical Devices official website — http://www.dunemedical.com